CLINICAL TRIAL: NCT05358119
Title: Characterising Musculoskeletal Pain in People Living With Long COVID - a Prospective Longitudinal Study
Brief Title: Musculoskeletal Pain in Long COVID
Acronym: MUSLOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: Leeds Comunity Healthcare NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Manoj Sivan, Associate Professor and Consultant in Rehabilitation Medicine, University of Leeds
Other Study IDs: 296125
Record Dates: First submitted 2022-04-30; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: COVID-19; Musculoskeletal Pain
MeSH Terms: conditions — COVID-19; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective cohort: Patients with long COVID and new-onset musculoskeletal pain

SUMMARY:
Long COVID is a new disease, with musculoskeletal pain being one of the common presenting symptoms. This longitudinal study will explore the long COVID musculoskeletal pain aetiology, pathophysiology, impact on function and quality of life, prognosis and its natural evolution.

DETAILED DESCRIPTION:
Long COVID is defined as signs and symptoms that develop during or after an infection consistent with COVID-19, continue for more than four weeks and are not explained by an alternative diagnosis. It has been estimated there are 2 million people in the UK alone with long COVID symptoms. Most people with long COVID experience some limitation to their daily activities. This causes new challenges to the patients and their families as well as to the healthcare system. Musculoskeletal (MSK) pain is one of the most common reported symptoms in long COVID. The causes and underlying mechanisms of MSK pain in long COVID are not fully understood yet. A few underlying mechanisms have been hypothesised to cause the pain including detrimental impacts of the virus on neurological functions and central nervous system; immunologic aberrations and inflammatory damage in response to the acute infection; expected sequelae of post-critical illness involving deconditioning process following a period of inactivity, bed rest or sedentary lifestyle associated with the viral infection.

The purpose of this study is to investigate the clinical characteristics, etiopathological mechanisms and the natural course of pain, and to understand its physical and psychosocial consequences. We will also analyse the correlation of pain to clusters of long COVID symptoms. We anticipate the results of this study will help the healthcare providers to deliver adequate management for patients with long COVID.

This is a longitudinal study to observe 100 patients with long COVID pain throughout an 18-month period. Pain assessment will be undertaken using validated methods, that include blood tests to detect inflammatory biomarkers, clinical examination, standardised pain instruments/scales, Quantitative Sensory Testing to measure changes in sensitivity, and electroencephalography to measure brain network activity. Physical activity measurements include Timed Up and Go Test to assess balance and mobility, Rated Perceived Exertion Scale to measure exercise intensity, and Hand-Grip Dynamometer test to measure handgrip strength. In addition, we will use psychological assessment tools to assess the severity of depression and anxiety, and self-efficacy and pain-related thoughts.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who have tested positive for COVID-19 or self-reported symptoms of COVID-19 confirmed by an independent clinician.
2. New onset musculoskeletal pain that develops during or following an infection consistent with COVID-19, continues for 4 weeks or more and is not explained by an alternative diagnosis.
3. Age 18 years or older.
4. Ability of participant to understand and the willingness to sign a written informed consent document.
5. Stated willingness to comply with all study procedures and availability for the duration of the study.
6. Ability of participant to read and understand English.

Exclusion Criteria:

1. People with pre-covid chronic pain syndrome.
2. Unable to provide informed consent.
3. Specific exclusion for Electroencephalogram (EEG): Patients with history of epileptic seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to recruit 100 individuals with new-onset musculoskeletal pain consistent with COVID-19.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory | 18 months
  It is an outcome measures pain severity, the impact of pain on daily function, the location of pain, pain medications and amount of pain relief in the past 24 hours of past week. It is originally developed to assess cancer pain but has been shown to have utility in chronic pain (Tan et al., 2004), with acceptable internal consistency (Cronbach α 0.85 intensity and 0.88 for interference) a stable 2-factor structure, and sensitivity to change with treatment. Similar qualities have been demonstrated in patients with musculoskeletal pain (Celik et al., 2016). There is no scoring algorithm for the Brief Pain Inventory, but "worst pain" or the arithmetic mean of four severity items can be used as measures of pain severity, and the arithmetic mean of the seven interference items can be used as a measure of pain interference.

SECONDARY OUTCOMES:
C19-YRS (Yorkshire Rehabilitation Scale) | 18 months
  C19-YRS (Yorkshire Rehabilitation Scale) is a Long COVID specific outcome measure developed by the CI (MS) and the Leeds Covid rehabilitation team. It gives a symptom severity score, functional disability score and overall health state score. It has been validated for use in Long COVID patients and has been shown to have good reliability. The scale will be used in this study to comprehensive measure the most relevant symptoms of Long COVID. This will allow us look at associations between MSK pain and other symptoms of Long COVID.
Patient Health Questionnaire-9 (PHQ-9) | 18 months
  The PHQ-9 is a screening instrument with 9 items, developed to measure depression. For each item the patients are asked to assess how much they were bothered by the symptoms over the last two weeks. There are four answer options: not at all (0), several days (1), more than half of the days (2), and nearly every day (3). The sum score (range 0 to 27) indicates the degree of depression, with scores of ≥5, ≥10, and ≥15 representing mild, moderate, and severe levels of depression.
EuroQol 5D (EQ-5D-5L) | 18 months
  The EQ-5D-5L is a widely used generic measure of health status consisting of two parts. The first part (the descriptive system) assesses health in five dimensions (MOBILITY, SELFCARE, USUAL ACTIVITIES, PAIN / DISCOMFORT, ANXIETY / DEPRESSION), each of which has five levels of response (no problems, slight problems, moderate problems, severe problems, and unable to). The second part of the EQ-5D questionnaire provides a descriptive profile that can be used to generate a health state profile. Health state index scores generally range from less than 0 (where 0 is a health state equivalent to death; negative values are valued as worse than death) to 1 (perfect health), with higher scores indicating higher health utility, though health state preferences can differ between countries. This part of the questionnaire consists of a VAS on which the patient rates his / her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
Blood inflammatory markers | 18 months
  Blood test known as 'inflammatory markers' can detect inflammation in the body, caused by many diseases including infections and auto-immune conditions. It helps to distinguish between inflammatory and noninflammatory causes of pain. The blood tests will be undertaken in this study to perform the measurements of serum inflammatory markers at baseline and follow-up visits. This measurement will include inflammatory markers such as: IL-1β, IL-6 and TNF-α.
Electroencephalogram sprectral analysis | 18 months
  It is an electrophysiological monitoring method to record electrical activity of the brain. It is typically non-invasive, with electrodes placed along the scalp. The procedure begins with the participant lying on the exam table or bed. The technician puts about 20 small sensors on the scalp. Theses sensors (electrodes) pick up electrical activity from neurons and send them back to a machine, they show up as series of lines records on paper or displayed on a computer screen. When recording begins, participants asked to remain still with their eyes open first, then with them closed
Quantitative sensory testing (QST) | 18 months
  QST systems have been developed to assess and quantify sensory function in patients with neurologic symptoms or in those at risk of developing neurologic disease. QST measures the detection threshold of accurately calibrated sensory stimuli. investigates the submodalities of the somatosensory system, such as temperature, touch, vibration, and pain. It provides information on the state of peripheral sensory nerves, as well as pain perception and central sensitization.
Timed Up and Go Test (TUG) | 18 months
  The timed up and go (TUG) is an outcome measure to assess balance and mobility. The TUG is recommended as a routine screening test for falls in guidelines published by the American Geriatric Society and the British Geriatric Society, and the National Institute of Clinical Evidence (NICE) guidelines also support use the TUG for assessment of gait and balance in the prevention of falls in older people. Participants start the test in a seated position, stand up upon a command to walk for 3 m, turn around and walk back to the chair and sit down. The participants supposed to complete this as quickly as possible, while being as comfortable and as safe as possible. A stopwatch measures the time (in seconds) above 12 second is considered as the cut-off.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Sivan, MD, Principal Investigator — University of Leeds
Locations (2):
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds, England
  - Leeds Community Healthcare NHS Trust, Leeds, England

IPD SHARING:
Plan to Share IPD: Undecided
This will be made available on request